CLINICAL TRIAL: NCT00852501
Title: Characterization of Receptors Present in Non-functioning Pituitary Macroadenomas by Reverse Transcriptase- Polymerase Chain Reaction (RT-PCR)
Brief Title: Characterization of Receptors in Non-functioning Pituitary Macroadenomas
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cook County Health (Other Government)
Collaborators: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Leon Fogelfeld, M.D., Cook County Health
Other Study IDs: 06-044
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Pituitary Tumor
Keywords: Non-functioning pituitary adenoma; RTPCR; Hormonal receptors
MeSH Terms: conditions — Pituitary Neoplasms | interventions — Reverse Transcriptase Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A small piece of the pituitary macradenoma removed at surgery will be frozen to perform RT-PCR
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Non-functioning pituitary macroadenoma: The performance of surgery is the standard of care in the management of non-functioning pituitary macroadenomas. The tissue obtained during surgery is routinely sent for histopathological examination. A piece of the tissue will undergo receptor characterisation via RT-PCR.
  Interventions: Other: To perform RT-PCR on the tissue obtained during surgery

INTERVENTIONS:
Other: To perform RT-PCR on the tissue obtained during surgery — The performance of surgery is the standard of care in the management of non-functioning pituitary macroadenomas. The tissue obtained during surgery is routinely sent for histopathological examination. A piece of the tissue will undergo receptor characterisation via RT-PCR.
  Other Names: Reverse Transcriptase polymerase chain reaction

SUMMARY:
Characterization of receptors present in non-functioning pituitary macroadenomas by Reverse Transcriptase- Polymerase Chain Reaction (RT-PCR) would assist with targeted medical therapy based on the information obtained by immunohistochemistry and RT-PCR.

DETAILED DESCRIPTION:
The pituitary gland in the brain is the master hormonal gland and is surrounded by important nerves and blood vessels. The pituitary gland can develop various types of tumors, some which do not produce any hormones and are called non-functioning pituitary adenomas. These non-functioning tumors can grow and can cause compression of these important structures. The usual treatment of large non-functioning pituitary macroadenoma is surgery. As it is surrounded by neuro-vascular bundles, this makes complete removal of the tumor sometimes impossible and even dangerous. A large number of subjects will still have some residual tumor post-surgery. The risks of residual tumor are further growth with compression and compromise of the function of surrounding vital organs especially vision.

If there is further growth of the tumor the options at present are repeat surgery or radiotherapy. Repeat surgery involves all the risks associated with brain surgery and sometimes may not be possible if very close to vital organs, while radiotherapy will over a period of time lead to complete or partial deficiency of pituitary hormone function and has been associated with long term cognitive deficits. In addition radiotherapy has a lag time of 12-24 months prior to onset of action.

However, pituitary tumors that do not actively secrete hormones may still harbour receptors to various hormones. The blockage of these receptors by various medications may enable us to stop the tumor from growing or recurring after surgery. This may open up a novel means of treatment of these non functioning tumors. So far there is very little information in the literature about the type of receptors present in these tumors.

Our study proposes to obtain a piece of the tissue removed during surgery and perform receptor characterization to help improve our knowledge in that area. Also correlating the receptor status with the clinical, hormonal and radiological profile of the patients may help to develop improved treatment strategies in the future and help us to predict the possibility of tumor regrowth.

ELIGIBILITY:
Inclusion Criteria:

1. Adults, both males and females age 18 years old or more
2. Pituitary tumor more than 10 mm in diameter diagnosed by MRI
3. No clinical or laboratory evidence of pituitary hormone oversecretion (non-functioning pituitary macroadenoma)

Exclusion Criteria:

1. Subjects with pituitary tumors less than 10 mm in diameter
2. Subjects with clinical or laboratory evidence of hormone oversecretion
3. Presence of dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects who are diagnosed with a non-functioning pituitary macroadenoma who are scheduled for surgery.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2006-03; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
To determine the expression of hormonal receptors in clinically non-functioning pituitary macroadenomas by RT - PCR and immunohistochemistry. | 2 years

SECONDARY OUTCOMES:
To correlate the clinical, hormonal and radiological characteristics of the patients with pituitary tumors with the hormonal receptors status. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ambika Babu, MD, Principal Investigator — Cook County Health
Locations (1):
- John H Stroger Jr. Hospital of Cook County, Chicago, Illinois, United States